CLINICAL TRIAL: NCT03015181
Title: VRC 605: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB075-00-AB (VRC07-523LS), Administered Intravenously or Subcutaneously to Healthy Adults
Brief Title: VRC 605: Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB075-00-AB (VRC07-523LS), Administered Intravenously or Subcutaneously to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 170030; 17-I-0030 (Other: NIH)
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: HIV Prevention
Keywords: Broadly Neutralizing; HIV Prevention; Anti-Drug Antibody; HIV-1; Immune Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1: 1 mg/kg IV Single Dose (Experimental): Group 1 subjects received a single IV infusion of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0 at a dose of 1 mg/kg.
  Interventions: Biological: VRC-HIVMAB075-00-AB
- Group 2: 5 mg/kg IV Single Dose (Experimental): Group 2 subjects received a single IV infusion of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0 at a dose of 5 mg/kg.
  Interventions: Biological: VRC-HIVMAB075-00-AB
- Group 3: 5 mg/kg SC Single Dose (Experimental): Group 3 subjects received a single SC injection of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0 at a dose of 5 mg/kg.
  Interventions: Biological: VRC-HIVMAB075-00-AB
- Group 4: 20 mg/kg IV Single Dose (Experimental): Group 4 subjects received a single IV infusion of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0 at a dose of 20 mg/kg.
  Interventions: Biological: VRC-HIVMAB075-00-AB
- Group 5: 40 mg/kg IV Single Dose (Experimental): Group 5 subjects received a single IV infusion of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0 at a dose of 40 mg/kg.
  Interventions: Biological: VRC-HIVMAB075-00-AB
- Group 6: 5 mg/kg SC Multiple Doses (Experimental): Group 6 subjects received a SC injection of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0, Week 12 and Week 24 at a dose of 5 mg/kg.
  Interventions: Biological: VRC-HIVMAB075-00-AB
- Group 7: 20 mg/kg IV Multiple Doses (Experimental): Group 7 subjects received an IV infusion of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0, Week 12 and Week 24 at a dose of 20 mg/kg.
  Interventions: Biological: VRC-HIVMAB075-00-AB

INTERVENTIONS:
Biological: VRC-HIVMAB075-00-AB — VRC07-523LS is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
  Other Names: VRC07-523LS

SUMMARY:
Background:

Human immunodeficiency virus (HIV) is a global health threat. The body uses antibodies to fight infection. VRC07-523LS is an antibody directed against HIV. It may be used to prevent mother-to-child transmission of HIV. It may also prevent sexual transmission of HIV and treat HIV-1 infected people.

Objective:

To test the safety, tolerability, dose, and pharmacokinetics of VRC07-523LS in healthy adults.

Eligibility:

Healthy people ages 18-50

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Participants will be assigned to 1 of 7 groups:

Groups 1-5 will get the drug at 1 visit and then be observed for 24 weeks.

Groups 6 and 7 will get the drug at 1 visit every 12 weeks, for a total of 3 doses over 48 weeks.

Participants will get the drug in 1 of 2 ways:

Infusion into a vein over at least 30 minutes. Participants will have blood tests 1, 3, and 6 hours after the infusion. They will have 1-3 visits during that week. Those in Group 7 will have 4-5 visits in the week after their second and third doses.

Injection into the fatty tissue under the skin. Participants will have blood tests before the injection. They will have 1-3 visits during that week. Those in Group 6 will have 4-5 visits after the second and third doses.

Visits include:

Physical exam

Blood and urine tests

Optional oral swabs to collect saliva

Participants will keep a diary of their temperature and symptoms for 3 days after each dose.

DETAILED DESCRIPTION:
This is the first study of the VRC-HIVMAB075-00-AB (VRC07-523LS) monoclonal antibody (MAb) in healthy adults. It is a phase 1, dose-escalation study to examine safety, tolerability, dose, and pharmacokinetics of VRC07-523LS. The hypothesis is that VRC07-523LS will be safe for administration to healthy adults by the intravenous (IV) and subcutaneous (SC) routes.

Healthy adults 18-50 years of age will be enrolled. There are 4 open-label, dose escalations of VRC07-523LS from 1 mg/kg IV to 40 mg/kg IV, 1 route escalation from IV to SC, and 2 open-label groups to assess repeat dosing. Groups 1-5 are expected to include 3 subjects and Groups 6-7 are expected to enroll 5 subjects. Subjects will be followed for 24 weeks after the last study product administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following criteria:

* Able and willing to complete the informed consent process.
* 18 to 50 years of age.
* Based on history and examination, must be in good general health and without history of any of the conditions listed in the exclusion criteria.
* Willing to have blood samples collected, stored indefinitely, and used for research purposes.
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
* Willing to adhere to reduced risk sexual behavior during study participation.
* Screening laboratory values within 84 days prior to enrollment must meet the following criteria:

  * White Blood Cell (WBC) 2,500-12,000/mm^3.
  * WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval.
  * Platelets = 125,000 - 400,000/mm^3.
  * Hemoglobin within institutional normal range.
  * Creatinine less than or equal to 1.1 x upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) less than or equal to 1.25 x ULN.
* Negative for HIV infection by the FDA approved method of detection.
* Female-Specific Criteria:

  * If a woman is of reproductive potential and sexually active with a male partner, then she agrees to use an effective means of birth control from the time of study enrollment until the last study visit, or to be monogamous with a partner who has had a vasectomy.
  * Negative Beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

* Previous receipt of licensed or investigational monoclonal antibody.
* Weight >115 kg.
* Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis prior to enrollment that has a reasonable risk of recurrence during the study.
* Hypertension that is not well controlled.
* Woman who is breast-feeding, or planning to become pregnant during the study participation.
* Receipt of any investigational study agent within 28 days prior to enrollment.
* Any other chronic or clinically significant medical condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer, including but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of: drug or alcohol abuse, asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Gaudinski, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudicell RS, Kwon YD, Ko SY, Pegu A, Louder MK, Georgiev IS, Wu X, Zhu J, Boyington JC, Chen X, Shi W, Yang ZY, Doria-Rose NA, McKee K, O'Dell S, Schmidt SD, Chuang GY, Druz A, Soto C, Yang Y, Zhang B, Zhou T, Todd JP, Lloyd KE, Eudailey J, Roberts KE, Donald BR, Bailer RT, Ledgerwood J; NISC Comparative Sequencing Program; Mullikin JC, Shapiro L, Koup RA, Graham BS, Nason MC, Connors M, Haynes BF, Rao SS, Roederer M, Kwong PD, Mascola JR, Nabel GJ. Enhanced potency of a broadly neutralizing HIV-1 antibody in vitro improves protection against lentiviral infection in vivo. J Virol. 2014 Nov;88(21):12669-82. doi: 10.1128/JVI.02213-14. Epub 2014 Aug 20. PMID 25142607
- [Background] Wu X, Yang ZY, Li Y, Hogerkorp CM, Schief WR, Seaman MS, Zhou T, Schmidt SD, Wu L, Xu L, Longo NS, McKee K, O'Dell S, Louder MK, Wycuff DL, Feng Y, Nason M, Doria-Rose N, Connors M, Kwong PD, Roederer M, Wyatt RT, Nabel GJ, Mascola JR. Rational design of envelope identifies broadly neutralizing human monoclonal antibodies to HIV-1. Science. 2010 Aug 13;329(5993):856-61. doi: 10.1126/science.1187659. Epub 2010 Jul 8. PMID 20616233
- [Result] Gaudinski MR, Houser KV, Doria-Rose NA, Chen GL, Rothwell RSS, Berkowitz N, Costner P, Holman LA, Gordon IJ, Hendel CS, Kaltovich F, Conan-Cibotti M, Gomez Lorenzo M, Carter C, Sitar S, Carlton K, Gall J, Laurencot C, Lin BC, Bailer RT, McDermott AB, Ko SY, Pegu A, Kwon YD, Kwong PD, Namboodiri AM, Pandey JP, Schwartz R, Arnold F, Hu Z, Zhang L, Huang Y, Koup RA, Capparelli EV, Graham BS, Mascola JR, Ledgerwood JE; VRC 605 study team. Safety and pharmacokinetics of broadly neutralising human monoclonal antibody VRC07-523LS in healthy adults: a phase 1 dose-escalation clinical trial. Lancet HIV. 2019 Oct;6(10):e667-e679. doi: 10.1016/S2352-3018(19)30181-X. Epub 2019 Aug 28. PMID 31473167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited at the NIH Clinical Center in Bethesda, Maryland.
Period: Overall Study
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses
Started | 4 | 3 | 3 | 3 | 3 | 5 | 5
Received VRC07-523LS Per Protocol | 3 | 3 | 3 | 3 | 3 | 4 | 4
Discontinued VRC07-523LS Administrations | 1 (One Group 1 subject decided not to receive the VRC07-523LS infusion) | 0 | 0 | 0 | 0 | 1 (One Group 6 subject received only 1 of 3 scheduled doses prior to withdrawing from the study) | 1 (One Group 7 subject received only 1 of 3 scheduled doses due to an unrelated intercurrent illness)
Completed | 3 | 3 | 3 | 3 | 3 | 4 (Group 6 subject who received only 1 dose chose to withdraw from study after the first administration) | 4 (Group 7 subject who received only 1 dose was withdrawn after unrelated intercurrent illness resolved)
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Enrolled, but product never administered | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 5 | 5 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (7.0) | 28.0 (9.5) | 30.0 (7.0) | 27.0 (2.6) | 40.0 (10.4) | 25.8 (4.1) | 30.0 (10.6) | 29.2 (8.1)
Age, Customized [Count of Participants; unit: Participants]
  21-30 years | 3 | 2 | 2 | 3 | 1 | 4 | 3 | 18
  31-40 years | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 5
  41-50 years | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 1 | 3 | 5 | 2 | 15
  Male | 2 | 1 | 3 | 2 | 0 | 0 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 4
  Not Hispanic or Latino | 4 | 3 | 2 | 2 | 2 | 4 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
  White | 2 | 2 | 2 | 2 | 1 | 4 | 3 | 16
  Multiracial | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 4
Weight [Mean (Standard Deviation); unit: kg] | 75.8 (4.6) | 65.5 (17.3) | 89.4 (15.0) | 75.9 (11.0) | 67.2 (20.1) | 55.2 (7.1) | 76.1 (11.4) | 71.3 (14.9)
Education [Count of Participants; unit: Participants]
  High school graduate/GeneralEducationalDevelopment | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  College/University | 2 | 2 | 2 | 2 | 2 | 4 | 4 | 18
  Advanced degree | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 3 Days of Any Product Administration
Description: Subjects recorded 3-day systemic symptoms in a diary after each study product administration. Solicited systemic symptoms include: unusually tired/feeling unwell, muscles aches, headache, chills, nausea, temperature and joint pain. Subjects recorded highest measured temperature daily. Clinicians reviewed the diary with the subject and collected resolution information for any symptoms that were not resolved within 3 days. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of subjects reporting any systemic symptom at the worst severity. Solicited reactogenicity was recorded without an attribution assessment. Grading was done by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0.
Time Frame: 3 days after each product administration
Population: Subjects who received VRC07-523LS (N=25), where "N" signifies number of subjects analyzed for this outcome measure. Groups 1, 2, 4, 5 and 7 are IV administration groups and Groups 3 and 6 are SC administration groups, with Groups 6 and 7 receiving multiple doses.
Measure: Count of Participants; unit: Participants
Groups:
- Group 7: 20 mg/kg IV Multiple Doses: Dose 1: Group 7 subjects who received an IV infusion of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0 at a dose of 20 mg/kg.
  VRC-HIVMAB075-00-AB: VRC07-523LS is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Group 7: 20 mg/kg IV Multiple Doses: Dose 2: Group 7 subjects who received an IV infusion of VRC07-523LS (VRC-HIVMAB075-00-AB) on Week 12 at a dose of 20 mg/kg.
  VRC-HIVMAB075-00-AB: VRC07-523LS is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Group 7: 20 mg/kg IV Multiple Doses: Dose 3: Group 7 subjects who received an IV infusion of VRC07-523LS (VRC-HIVMAB075-00-AB) on Week 24 at a dose of 20 mg/kg.
  VRC-HIVMAB075-00-AB: VRC07-523LS is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Overall IV Groups: Total number of subjects who received an IV infusion of VRC07-523LS (VRC-HIVMAB075-00-AB) - Groups 1, 2, 4, 5 and 7 are IV administration groups
- Group 6: 5 mg/kg SC Multiple Doses: Dose 1: Group 6 subjects who received a SC injection of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0 at a dose of 5 mg/kg.
  VRC-HIVMAB075-00-AB: VRC07-523LS is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Group 6: 5 mg/kg SC Multiple Doses: Dose 2: Group 6 subjects who received a SC injection of VRC07-523LS (VRC-HIVMAB075-00-AB) on Week 12 at a dose of 5 mg/kg.
  VRC-HIVMAB075-00-AB: VRC07-523LS is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Group 6: 5 mg/kg SC Multiple Doses: Dose 3: Group 6 subjects who received a SC injection of VRC07-523LS (VRC-HIVMAB075-00-AB) on Week 24 at a dose of 5 mg/kg.
  VRC-HIVMAB075-00-AB: VRC07-523LS is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Overall SC Groups: Total number of subjects who received an SC injection of VRC07-523LS (VRC-HIVMAB075-00-AB) - Groups 3 and 6 are SC administration groups
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 7: 20 mg/kg IV Multiple Doses: Dose 1 | Group 7: 20 mg/kg IV Multiple Doses: Dose 2 | Group 7: 20 mg/kg IV Multiple Doses: Dose 3 | Overall IV Groups | Group 3: 5 mg/kg SC Single Dose | Group 6: 5 mg/kg SC Multiple Doses: Dose 1 | Group 6: 5 mg/kg SC Multiple Doses: Dose 2 | Group 6: 5 mg/kg SC Multiple Doses: Dose 3 | Overall SC Groups
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 4 | 17 | 3 | 5 | 4 | 4 | 8
Participants
  Malaise: None | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 14 | 3 | 2 | 4 | 4 | 5
  Malaise: Mild | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 3 | 0 | 0 | 3
  Malaise: Moderate | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 3 | 2 | 3 | 2 | 4 | 3 | 3 | 14 | 3 | 3 | 4 | 4 | 6
  Myalgia: Mild | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 2
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Headache: None | 3 | 3 | 3 | 2 | 4 | 3 | 4 | 15 | 3 | 3 | 3 | 4 | 5
  Headache: Mild | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 3
  Headache: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 3 | 3 | 3 | 2 | 4 | 3 | 3 | 15 | 3 | 4 | 4 | 4 | 7
  Chills: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Chills: Moderate | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 3 | 3 | 3 | 2 | 5 | 4 | 4 | 16 | 3 | 4 | 4 | 4 | 7
  Nausea: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Nausea: Moderate | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 16 | 3 | 5 | 4 | 4 | 8
  Temperature: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 3 | 3 | 3 | 2 | 5 | 4 | 3 | 15 | 3 | 3 | 4 | 4 | 6
  Joint Pain: Mild | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom Reported: None | 3 | 2 | 3 | 2 | 3 | 3 | 3 | 13 | 3 | 1 | 3 | 4 | 3
  Any Systemic Symptom Reported: Mild | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 4 | 1 | 0 | 5
  Any Systemic Symptom Reported: Moderate | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Any Product Administration
Description: Local symptoms assessed and recorded by the clinicians. Solicited local symptoms include pain/tenderness, swelling, redness, bruising, and pruritus (itchiness) at the product administration site. Clinicians assessed the study product administration site for local symptoms on the day of product administration after completion of the administration and on Days 1, 2 and 7 post administration. Subjects were counted once for each symptom at the worst severity if they experienced the symptom at any severity during the reporting period. If symptoms were experienced, clinicians collected resolution information for any symptom that was not resolved within 7 days. The number reported for "Any Local Symptom" is the number of subjects reporting any local symptom at the worst severity. Solicited reactogenicity recorded without an attribution assessment. If symptoms were reported, grading was done by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0.
Time Frame: 7 days after each product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Group 6: 5 mg/kg SC Multiple Doses: Dose 1: Group 6 subjects received a SC injection of VRC07-523LS (VRC-HIVMAB075-00-AB) on Day 0 at a dose of 5 mg/kg.
  VRC-HIVMAB075-00-AB: VRC07-523LS is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 7: 20 mg/kg IV Multiple Doses: Dose 1 | Group 7: 20 mg/kg IV Multiple Doses: Dose 2 | Group 7: 20 mg/kg IV Multiple Doses: Dose 3 | Overall IV Groups | Group 3: 5 mg/kg SC Single Dose | Group 6: 5 mg/kg SC Multiple Doses: Dose 1 | Group 6: 5 mg/kg SC Multiple Doses: Dose 2 | Group 6: 5 mg/kg SC Multiple Doses: Dose 3 | Overall SC Groups
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 4 | 17 | 3 | 5 | 4 | 4 | 8
Participants
  Pain/Tenderness: None | 3 | 3 | 2 | 3 | 5 | 4 | 4 | 16 | 2 | 2 | 1 | 2 | 4
  Pain/Tenderness: Mild | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 2 | 4
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: None | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 16 | 3 | 5 | 4 | 4 | 8
  Bruising: Mild | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Bruising: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 3 | 3 | 3 | 3 | 5 | 4 | 4 | 17 | 3 | 5 | 4 | 4 | 8
  Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 3 | 3 | 3 | 3 | 5 | 4 | 4 | 17 | 3 | 5 | 4 | 3 | 7
  Redness: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Pruritus: None | 3 | 3 | 3 | 3 | 5 | 4 | 4 | 17 | 3 | 5 | 4 | 4 | 8
  Pruritus: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritus: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom Reported: None | 3 | 3 | 2 | 3 | 4 | 4 | 4 | 15 | 2 | 2 | 1 | 1 | 4
  Any Local Symptom Reported: Mild | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 3 | 2 | 3
  Any Local Symptom Reported: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

3. Primary Outcome: Number of Subjects Reporting 1 or More Unsolicited Non-Serious Adverse Events
Description: Unsolicited adverse events (AEs) collected during the period from study product administration at Day 0 through 56 days after the last product administration. After the indicated time period through the last expected study visit at 24 weeks after the last product administration, only new chronic medical conditions collected as unsolicited AEs. The number reported is the number of subjects who experienced at least one AE in the reporting period. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Through 24 weeks after the last product administration
Population: Subjects who received VRC07-523LS (N=25), where "N" signifies number of subjects analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Total number of subjects who received VRC07-523LS (VRC-HIVMAB075-00-AB)
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses | Overall
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 5 | 25
Participants
  Related to study product | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 4
  Unrelated to study product | 2 | 1 | 1 | 0 | 0 | 5 | 3 | 12

4. Primary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events (SAEs) collected during the period from study product administration at Day 0 through 24 weeks after the last product administration.
Time Frame: Through 24 weeks after the last product administration
Population: Subjects who received VRC07-523LS (N=25), where "N" signifies number of subjects analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses | Overall
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 5 | 25
Participants
  Related to study product | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unrelated to study product | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of VRC07-523LS: Single Dose Groups
Description: Cmax is the peak serum concentration that VRC07-523LS achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group.
  Serum was collected at the following time points:
  Groups 1, 2, 4, and 5: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hours post infusion, followed by Weeks 1-4, 8, 12, 16, 20, and 24 post infusion; Group 3: Pre-injection (baseline) and 24, 48, 72 hours post injection, and Weeks 1-4, 8, 12, 16, 20, and 24 post injection
Time Frame: Up to 24 weeks post product administration
Population: Pharmacokinetic (PK) parameters shown for all subjects who received at least one administration of VRC07-523LS, and represents the first dose only. One subject in Group 7 (multiple doses at 20 mg/kg IV) who only received a single dose was analyzed with Group 4 (single dose at 20 mg/kg IV).
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3
µg/mL | 47 (16) | 240 (35) | 50 (11) | 869 (190) | 1630 (644)

6. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of VRC07-523LS: Multiple Dose Groups
Description: Cmax is the peak serum concentration that VRC07-523LS achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group.
  Serum was collected at the following time points for Groups 6 and 7 after Dose 1 and Dose 3:
  Group 6, Dose 1: Pre-injection (baseline) and 24, 48, and 72 hours post injection, followed by Weeks 1, 2, 4 and 8 post injection; Group 6, Dose 3: Pre-injection (Week 24) and 72 hours post injection, followed by Weeks 25-28 and every 4 weeks up to 48 weeks post injection; Group 7, Dose 1: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hrs post infusion, followed by Weeks 1, 2, 4 and 8 post infusion; Group 7, Dose 3: Pre-infusion (Week 24), end of infusion and 1 hour post infusion followed by Weeks 25-28 and every 4 weeks up to 48 weeks post infusion
Time Frame: Through 24 weeks after the last product administration
Population: Pharmacokinetic (PK) parameters shown for all subjects who received at least one administration of VRC07-523LS, and represents the first dose only. One subject in Group 7 (multiple doses at 20 mg/kg IV) who only received a single dose was analyzed with Group 4 (single dose at 20 mg/kg IV). For Dose 3, values calculated from 4 subjects per group.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses
Number analyzed (Participants) | 5 | 4
µg/mL
  Dose 1 | 38 (17) | 1196 (74)
  Dose 3: number analyzed (Participants) | 4 | 4
  Dose 3 | 37 (12) | 799 (98)

7. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of VRC07-523LS
Description: Tmax is the time it takes to reach Cmax of VRC07-523LS after it has been administered; it is determined based on the summary PK curve for each study group
  Serum was collected at the following time points:
  Groups 1, 2, 4, and 5: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hours post infusion, followed by Weeks 1-4, 8, 12, 16, 20, and 24 post infusion; Group 3: Pre-injection (baseline) and 24, 48, 72 hours post injection, and Weeks 1-4, 8, 12, 16, 20, and 24 post injection; Group 6, Dose 1: Pre-injection (baseline) and 24, 48, and 72 hours post injection, followed by Weeks 1, 2, 4 and 8 post injection; Group 7, Dose 1: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hours post infusion, followed by Weeks 1, 2, 4 and 8 post infusion
Time Frame: Through 24 weeks after the last product administration for Groups 1-5 and through 8 weeks after the last product administration for Groups 6 and 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 5 | 4
days | 0.7 (0.5) | 0.04 (0.02) | 10 (9.5) | 0.3 (0.4) | 0.04 (0.02) | 5.7 (5.0) | 0.04 (0.02)

8. Secondary Outcome: 4 Week Mean Serum Concentration of VRC07-523LS
Description: The mean of individual subject VRC07-523LS serum concentrations by administered dose group
Time Frame: Week 4 post product administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 5 | 4
µg/mL | 14 (7.5) | 57 (11) | 31 (11) | 148 (28) | 272 (52) | 25 (13) | 242 (51)

9. Secondary Outcome: 12 Week Mean Serum Concentration of VRC07-523LS: Single Dose Groups
Description: The mean of individual subject VRC07-523LS serum concentrations by administered dose group
Time Frame: Week 12 post product administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3
µg/mL | 3.8 (0.7) | 57 (11) | 7.1 (1.3) | 44 (14) | 85 (30)

10. Secondary Outcome: 12 Week Mean Serum Concentration of VRC07-523LS: Multiple Dose Groups
Description: The mean of individual subject VRC07-523LS serum concentrations by administered dose group
Time Frame: Up to 12 weeks after each product administration
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses
Number analyzed (Participants) | 5 | 4
µg/mL
  Dose 1 | 6.3 (1.5) | 46 (13)
  Dose 3: number analyzed (Participants) | 4 | 4
  Dose 3 | 9.8 (2.5) | 71 (29)

11. Secondary Outcome: Area Under the Curve (AUC(0-inf)): Single Dose Groups
Description: The total area under the curve (AUC(inf)) was taken as the sum of the observed AUC up to the final concentration (AUC(obs)) plus the AUC after the final concentration (AUC(Clast-inf)) where AUC(Clast-inf) was estimated as Clast/lz.
  Serum was collected at the following time points:
  Groups 1, 2, 4, and 5: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hours post infusion, followed by Weeks 1-4, 8, 12, 16, 20, and 24 post infusion; Group 3: Pre-injection (baseline) and 24, 48, 72 hours post injection, and Weeks 1-4, 8, 12, 16, 20, and 24 post injection
Time Frame: Administration (0h) to 24 weeks post product administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg*d/mL
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3
µg*d/mL | 1381 (325) | 4551 (904) | 2189 (309) | 13748 (1853) | 25517 (5097)

12. Secondary Outcome: Area Under the Curve (AUC0-84D): Multiple Dose Groups
Description: The AUC0-84D represents the total drug exposure in 84 days after VRC07-523LS administration; it is determined based on the summary PK curve for each group.
  Serum was collected at the following time points for Groups 6 and 7 after Dose 1 and Dose 3:
  Group 6, Dose 1: Pre-injection (baseline) and 24, 48, and 72 hours post injection, followed by Weeks 1, 2, 4 and 8 post injection; Group 6, Dose 3: Pre-injection (Week 24) and 72 hours post injection, followed by Weeks 25-28 and every 4 weeks up to 48 weeks post injection; Group 7, Dose 1: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hrs post infusion, followed by Weeks 1, 2, 4 and 8 post infusion; Group 7, Dose 3: Pre-infusion (Week 24), end of infusion and 1 hour post infusion followed by Weeks 25-28 and every 4 weeks up to 48 weeks post infusion
Time Frame: Administration (0h) up to 84 days after each product administration
Population: Pharmacokinetic (PK) parameters shown for all subjects who received at least one administration of VRC07-523LS, and represents the first dose only. One subject in Group 7 (multiple doses at 20 mg/kg IV) who only received a single dose was analyzed with Group 4 (single dose at 20 mg/kg IV). For Dose 3, value calculated from 4 subjects per group.
Measure: Mean (Standard Deviation); unit: µg*d/mL
Arm/Group | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses
Number analyzed (Participants) | 5 | 4
µg*d/mL
  Dose 1 | 1440 (563) | 14760 (2646)
  Dose 3: number analyzed (Participants) | 4 | 4
  Dose 3 | 1671 (443) | 13573 (1115)

13. Secondary Outcome: VRC07-523LS Clearance Rate
Description: Rate of VRC07-523LS elimination divided by the plasma VRC07-523LS concentration; determined based on the summary PK curve for each study group.
  Serum was collected at the following time points:
  Groups 1, 2, 4, and 5: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hours post infusion, followed by Weeks 1-4 post infusion; Group 3: Pre-injection (baseline) and 24, 48, 72 hours post injection, and Weeks 1-4 post injection; Group 6, Dose 1: Pre-injection (baseline) and 24, 48, and 72 hours post injection, followed by Weeks 1, 2 and 4 post injection; Group 7, Dose 1: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hours post infusion, followed by Weeks 1, 2 and 4 post infusion
Time Frame: Administration (0h) to 28 days post product administration
Population: Pharmacokinetic (PK) parameters shown for all subjects who received at least one administration of VRC07-523LS. One subject in Group 7 (multiple doses at 20 mg/kg IV) who only received a single dose was analyzed with Group 4 (single dose at 20 mg/kg IV). Value following SC administration represents CL/F (apparent clearance).
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 7: 20 mg/kg IV Multiple Doses | Overall IV Groups | Group 3: 5 mg/kg SC Single Dose | Group 6: 5 mg/kg SC Multiple Doses | Overall SC Groups
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 17 | 3 | 5 | 8
mL/day | 70 (20) | 78 (18) | 110 (19) | 105 (14) | 101 (15) | 94 (22) | 226 (54) | 158 (34) | 184 (52)

14. Secondary Outcome: Overall IV Half-life (T1/2) of VRC07-523LS
Description: Half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
  Serum was collected at the following time points:
  Groups 1, 2, 4, and 5: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hours post infusion, followed by Weeks 1-4 and 8 post infusion; Group 3: Pre-injection (baseline) and 24, 48, 72 hours post injection, and Weeks 1-4 and 8 post injection; Group 6, Dose 1: Pre-injection (baseline) and 24, 48, and 72 hours post injection, followed by Weeks 1, 2, 4 and 8 post injection; Group 7, Dose 1: Pre-infusion (baseline), end of infusion (0h) and 1, 3, 6, 24 and 48 hours post infusion, followed by Weeks 1, 2, 4 and 8 post infusion
Time Frame: Administration (0h) to 56 days post product administration
Population: Pharmacokinetic (PK) parameters shown for all subjects who received at least one administration of VRC07-523LS. One subject in Group 7 (multiple doses at 20 mg/kg IV) who only received a single dose was analyzed with Group 4 (single dose at 20 mg/kg IV).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 7: 20 mg/kg IV Multiple Doses | Overall IV Groups | Group 3: 5 mg/kg SC Single Dose | Group 6: 5 mg/kg SC Multiple Doses | Overall SC Groups
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 17 | 3 | 5 | 8
days | 48 (26) | 32 (1.1) | 45 (5.2) | 42 (5.1) | 27 (1.8) | 38 (12) | 36 (6.7) | 31 (10) | 33 (8.9)

15. Secondary Outcome: Number of Single Dose Subjects Who Produced Anti-Drug Antibodies to VRC07-523LS
Description: Serum samples collected 4 weeks and 8 weeks after VRC07-523LS administration
Time Frame: Weeks 4 and 8 post product administration
Population: Subjects who received a single dose of VRC07-523LS via SC or IV administration. One subject in Group 7 (multiple doses at 20 mg/kg IV) who only received a single dose was analyzed with Group 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 3: 5 mg/kg SC Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 3
Participants
  Week 4: Subjects with Anti-Drug Antibodies | 0 | 0 | 0 | 0 | 0
  Week 8: Subjects with Anti-Drug Antibodies | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Multiple Dose Subjects Who Produced Anti-Drug Antibodies to VRC07-523LS
Description: Serum samples collected 4 weeks, 28 weeks and 32 weeks after VRC07-523LS administration
Time Frame: Weeks 4, 28 and 32 after the first product administration
Population: Subjects who received multiple doses of VRC07-523LS via SC or IV administration. One subject in Group 7 who only received a single dose was not included in this analysis but was analyzed with Group 4 (single dose at 20 mg/kg IV).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 6: 5 mg/kg SC Multiple Doses | Group 7: 20 mg/kg IV Multiple Doses
Number analyzed (Participants) | 5 | 4
Participants
  Week 4: Subjects with Anti-Drug Antibodies | 0 | 0
  Week 28: Subjects with Anti-Drug Antibodies | 0 | 0
  Week 32: Subjects with Anti-Drug Antibodies | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) included systemic AEs reported by subjects at the worst severity through 3 days post any product administration; and local administration site AEs reported for subjects at the worst severity through 7 days post any product administration. Unsolicited AEs were reported from the date of product administration through 56 days thereafter, and new chronic medical conditions and SAEs with onset any time following the date of last product administration through 24 weeks.
Description: Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of subjects reporting the event. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: 1 mg/kg IV Single Dose | Group 2: 5 mg/kg IV Single Dose | Group 4: 20 mg/kg IV Single Dose | Group 5: 40 mg/kg IV Single Dose | Group 7: 20 mg/kg IV Multiple Doses | Group 3: 5 mg/kg SC Single Dose | Group 6: 5 mg/kg SC Multiple Doses
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 1/3 | 2/3 | 5/5 | 2/3 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 1 mg/kg IV Single Dose (N=3) | Group 2: 5 mg/kg IV Single Dose (N=3) | Group 4: 20 mg/kg IV Single Dose (N=3) | Group 5: 40 mg/kg IV Single Dose (N=3) | Group 7: 20 mg/kg IV Multiple Doses (N=5) | Group 3: 5 mg/kg SC Single Dose (N=3) | Group 6: 5 mg/kg SC Multiple Doses (N=5)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 3
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Administration site pain/tenderness (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 3
Administration site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Administration site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Redness
Malaise (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Temperature (Fever)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 — Joint Pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT03015181/Prot_SAP_ICF_001.pdf